CLINICAL TRIAL: NCT04479618
Title: A Test of the Safety, Effectiveness, and Acceptability of an Improvised Dressing for Sickle Cell Leg Ulcers in a Tropical Climate
Brief Title: Test of the Safety, Effectiveness, & Acceptability of An Improvised Dressing for Sickle Cell Leg Ulcers in the Tropics
Acronym: SCLUJamaica
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benskin, Linda, PhD, RN, SRN (Ghana), CWCN, CWS, DAPWCA (Other)
Collaborators: Wound Healing Foundation (Other); University Hospital of the West Indies (Other); The University of The West Indies (Other); Ferris Mfg. Corp. (Industry)
Responsible Party: Principal Investigator, Linda Benskin, Principle investigator, Benskin, Linda, PhD, RN, SRN (Ghana), CWCN, CWS, DAPWCA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCLUJamaica2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sickle Cell Leg Ulcer
Keywords: sickle cell; chronic wounds; lower leg ulcer; venous ulcer; dressings, occlusive; sickle cell leg ulcer; dressings; bandages
MeSH Terms: conditions — Varicose Ulcer; Bites and Stings

STUDY DESIGN:
Intervention Model Description: A targeted-blinded, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: off-site wound experts and the local physicians verifying wound closure and/or complications will be blinded to the randomization group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Usual practice (negative control) (Active Comparator): After a member of the UHWI surgical team performs the initial cleansing/debriding, the control group (1) will have their ulcer dressed as usually done at UHWI. Wounds are dressed with saline-soaked gauze, covered with dry gauze. One wrap of stretch gauze will hold the dressing in place. Patients will clean the wound by vigorously wiping with gauze soaked in homemade normal saline (1 tsp salt/500ml water bottle), center to edges, at each dressing change, unless already very clean. Clean wounds will simply be irrigated with normal saline at each dressing change. Patients experienced with using papaya for debridement of their ulcers may apply it only to the open wound, avoiding contact with the periwound, to remove slough or eschar. If patients observe green exudate, they are permitted to add one teaspoon of vinegar to their bottle of saline. Dressings in group (1) will be changed daily. The dressings will be soaked off if they become adherent.
  Interventions: Device: Usual Practice
- improvised dressings (experimental) (Experimental): After initial cleansing/debriding, patients in the improvised dressing group (2) will then have a thin layer zinc oxide paste applied to the dried periwound, carefully avoiding the open wound. A piece of a clean new plastic bag (food-grade World Star 1 mil LD bags, or the equivalent, purchased from the Papine Market across John Golding Road from the University of the West Indies), cut slightly larger than the ulcer will be gently conformed to the moist wound contours and sealed onto the zinc oxide paste. The bag will be fenestrated with a small slit using a number 11 scalpel or clean scissors prior to placing it on the ulcer in order to allow excess fluid to escape. The edges of the slit will be approximated. Clean gauze will be placed lightly over the slit to capture escaping fluid. One wrap of stretch gauze will hold the dressing in place. Patients will be instructed to change the dressings daily, irrigating with normal saline at each dressing change.
  Interventions: Device: Improvised dressing
- advanced dressings (positive control) (Active Comparator): After initial cleansing/debriding, the advanced dressing group (3) will have a cut piece of a 4"x24" standard (pink) polymeric membrane dressing roll large enough to extend at least 0.5 cm beyond all open and closed (inflamed or damaged) wound edges applied as per the Instructions for Use (the periwound is blotted dry, but the wound bed remains moist from the final saline rinse). One wrap of stretch gauze will hold the polymeric membrane dressing in place. The approximate open wound edges will be marked on the dressing backing. As per the manufacturer's instructions for use, patients will change the dressings when saturation reaches any of the wound edges, as indicated by a change in color on the backing of the dressing, visible through the stretch gauze. Routine rinsing will not be performed; the wounds will be rinsed at dressing changes only if visible loose debris is present.
  Interventions: Device: Advanced dressing

INTERVENTIONS:
Device: Usual Practice — A saline soaked piece of gauze, conformed to the size of the open ulcer area, will be placed over the ulcer and held in place with a wrap of stretch gauze. Ulcers will be rinsed with saline at daily dressing changes, which will be conducted by the patient after they master the procedure.
  Other Names: Saline Gauze
  Arms: Usual practice (negative control)
Device: Improvised dressing — A piece of a new food-grade plastic bag, cut slightly larger than the ulcer, will be placed over the ulcer, sealed at the edges with an emollient to create an occlusive dressing. The dressing will be gently conformed to the ulcer contours to eliminate dead space, and a slit will be cut in the center to allow excess fluid to escape into a clean absorbent material placed over the slit. The device will be held in place with a wrap of stretch gauze. Ulcers will be rinsed with saline at daily dressing changes, which will be conducted by the patient after they master the procedure.
  Other Names: Wrap Therapy (modified for a tropical environment)
  Arms: improvised dressings (experimental)
Device: Advanced dressing — A piece of polymeric membrane dressing, cut to extend at least 0.5cm beyond the open ulcer edges, will be placed over the ulcer and held in place with a wrap of stretch gauze. The approximate wound edges will be marked on the back of the dressing. Dressing changes will consist only of removing the dressing when the saturation level, visible through the wound backing, reaches the mark indicating the dressing edges and applying a new cut dressing. Changes will be conducted by the patient after they master the procedure.
  Other Names: Polymeric membrane dressings; PolyMem
  Arms: advanced dressings (positive control)

SUMMARY:
One in 300 Jamaicans have HbSS sickle cell disease, and of these, up to 70% will suffer from sickle cell leg ulcers (SCLUs). Of these, 24% will have a chronic SCLU (one lasting longer than 6 months). SCLUs heal very slowly, and sometimes they never close. SCLU patients would benefit from an economical, less painful, dressing option. In addition, because SCLUs often compromise education and employment opportunities, improving wound care for this population benefits their entire community.

This three-armed evaluator-blinded randomized controlled trial will determine if a cut-to-fit food-grade plastic-based improvised dressing decreases pain, improves quality of life, and is safe, effective, and acceptable for managing SCLUs in Jamaica. The negative control will be usual practice, and the positive control will be the advanced wound dressing with the strongest evidence supporting its use in a tropical climate (polymeric membrane dressing).

Patients with SCLUs will be actively recruited from three adjacent parishes. The first 120 SCLU patients meeting study criteria presenting to UHWI, Mona, will be randomized immediately after initial cleansing/debriding into group (1) current usual practice, group (2) improvised dressings, or group (3) advanced dressings. Data will be added to each participant's data collection tool weekly. Results will be reported using descriptive statistics and ANCOVA. The expected outcome is both improvised and advanced dressing superiority to usual practice.

Because proposed improvised dressing materials are easily obtainable, their use would increase the capacity of wound patients to safely and effectively care for themselves.

Signed informed consent will be obtained from patients/parents. Only principal research investigators will have access to participant confidential information. The literature review demonstrates that risks are not higher than usual practice.

DETAILED DESCRIPTION:
This study's primary purpose is to determine if an improvised dressing, made from inexpensive materials available for purchase in rural as well as urban settings, is a safe and effective, culturally and medically acceptable choice for managing sickle cell leg ulcers in a tropical climate. Three research questions will be addressed:

1. Is the improvised dressing, consisting of a cut-to-fit new plastic bag sealed at the periwound with zinc oxide paste, safe and effective (see definitions, below) when compared with usual practice (saline-soaked gauze) and when compared with an advanced wound dressing (PMD), on sickle cell leg ulcers (SCLUs) in Jamaica?
2. Does use of the improvised dressing, when compared with usual practice, improve the quality of life of patients (decrease pain, increase ability to engage in desirable activities, decrease wound-related materials costs, decrease time required to perform dressing changes, improve Wound QoL scores, and improve ASCQ-Me pencil-and-paper interview scores) with SCLUs in Jamaica?
3. Is the improvised dressing culturally acceptable to health care providers, patients, and families for managing SCLUs in Jamaica?

The expected study outcome is improvised dressing superior effectiveness and quality of life, when compared with usual practice, without increased safety and acceptability issues. The improvised dressing is likely to be the least expensive choice, with the added benefit of being available as first aid treatment throughout Jamaica. The advanced dressing is likely to be more expensive with respect to materials costs, although fewer dressing changes are anticipated and pain medication expenses are likely to be reduced. Based upon the review of the literature, no serious infections or other safety issues are anticipated for any group. However, to ensure that complications are not overlooked, in addition to the onsite researchers' vigilance, weekly wound photos will be assessed for complications (signs of infection, wound deterioration, or clinically relevant maceration) by two off-site blinded wound experts.

Definitions:

Sickle cell leg ulcer - a wound in a HbSS or HbSβ0 positive patient, open greater than one month, below the level of the knee excluding the plantar surface of the foot.

Closed wound - 100% epithelialized with no discernible scab or exudate production (paper napkin remains dry when lightly pressed against area, and no recurrence in the subsequent two weeks)

Safe - infection and other complications (healing-impairing maceration, keloid, and contracture rates) not statistically significantly higher than usual practice, with no major adverse events attributable to the method

Effective - ulcer closure rates or ulcer surface area reduction rates not statistically significantly lower than usual practice

Acceptable - average acceptability scores of 4 or higher on a 1 - 5 scale

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HbSS or HbSβ0 sickle cell disease
* Ages 13 - 70 years at study initiation (able to comprehend and give consent)
* Males and females, pregnancy is not an issue
* Open wound below the knee, not including the plantar surface of the foot
* Wound open for longer than one month (defined as a chronic SCLU)
* Traumatic, spontaneous, or recurrent SCLU (all etiologies)

Exclusion Criteria:

* Patient younger than 13 years of age at study initiation
* Patient older than 70 years of age at study initiation
* Wound open for less than one month by conclusion of study enrollment period (acute wounds could be traumatic wounds unrelated to sickle cell diagnosis)
* Diagnosis of cancer, hypertension, or chronic renal failure
* Diabetes (will screen for undiagnosed diabetes)
* Active wound infection (evidenced by clinical signs of malodor, dark-colored or thick drainage, or significantly increased warmth at the periwound) which is not resolved by the conclusion of the study enrollment period
* Osteomyelitis (if osteomyelitis is suspected, an ESR will be drawn; > 70mm/h with high platelet levels and low serum albumin warrants a bone biopsy)
* Hydroxyurea use (may be a confound because it reduces inflammation and negates much of the pathology of SSD - may choose to abstain for the study)

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Benskin, PhD, Principal Investigator — Independent Nurse Researcher for Rural Tropical Areas, AND Ferris Mfg. Corp.; Rajeev Venugopal, MBBS, Study Chair — Consultant Plastic Surgeon, University Hospital of the West Indies
Locations (1):
- University Hospital of the West Indies, Mona, Kingston, Jamaica

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheet with de-identified data will be available upon request (by emailing the investigators)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study results have been published, for 10 years
Access Criteria: all interested parties

REFERENCES:
- [Background] Benskin LL. A review of the literature informing affordable, available wound management choices for rural areas of tropical developing countries. Ostomy Wound Manage. 2013 Oct;59(10):20-41. PMID 24106254
- [Background] Benskin LLL. Discovering the Current Wound Management Practices of Rural Africans [Dissertation]. 2013. Available from: http://utmb-ir.tdl.org/handle/2152.3/538
- [Derived] Scientific and Clinical Abstracts From WOCNext(R) 2022: Fort Worth, Texas diamond June 5-8, 2022. J Wound Ostomy Continence Nurs. 2022 May-Jun 01;49(3 Suppl 1):S1-S99. doi: 10.1097/WON.0000000000000882. No abstract available. PMID 35639023
- See also: Update on improvised dressings project as of May 2019 — http://rgdoi.net/10.13140/RG.2.2.28503.14247
- See also: Preliminary results to be presented at NCCHC 2023 — http://www.researchgate.net/publication/365368629

RESULTS

PARTICIPANT FLOW:
Groups:
- Improvised Dressings (Experimental): After initial cleansing/debriding, patients in the improvised dressing group (2) will then have a thin layer zinc oxide paste applied to the dried periwound, carefully avoiding the open wound. A piece of a clean new plastic bag (food-grade World Star 1 mil LD bags, or the equivalent, ...cut slightly larger than the ulcer will be gently conformed to the moist wound contours and sealed onto the zinc oxide paste. The bag will be fenestrated with a small slit using a number 11 scalpel or clean scissors prior to placing it on the ulcer in order to allow excess fluid to escape. The edges of the slit will be approximated. Clean gauze will be placed lightly over the slit to capture escaping fluid. One wrap of stretch gauze will hold the dressing in place. Patients will be instructed to change the dressings daily, irrigating with normal saline at each dressing change.
  Improvised dressing: A piece of a new food-grade plastic bag, cut slightly larger than the ulcer, will be placed over the ulcer, sealed at the edges with an emollient to create an occlusive dressing. The dressing will be gently conformed to the ulcer contours to eliminate dead space, and a slit will be cut in the center to allow excess fluid to escape into a clean absorbent material placed over the slit. The device will be held in place with a wrap of stretch gauze. Ulcers will be rinsed with saline at daily dressing changes, which will be conducted by the patient after they master the procedure.
Period: Overall Study
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Started | 18 | 14 | 16
Completed | 16 | 13 | 11
Not Completed | 2 | 1 | 5
Not completed — Agreed to randomization, but withdrew when it did not lead to assignment to Group 2 | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — No reliable phone and unable to come in weekly | 0 | 1 | 1
Not completed — Unable to comply with protocol due to physical disability plus social isolation (no assistance) | 0 | 0 | 1
Not completed — Intellectually disabled; caregivers neglected to follow protocol | 0 | 0 | 1
Not completed — Emotionally unstable; (e.g.,data unreliable - completed four weeks' forms on day they were received) | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Improvised Dressings (Experimental): After initial cleansing/debriding, patients in the improvised dressing group (2) will then have a thin layer zinc oxide paste applied to the dried periwound, carefully avoiding the open wound. A piece of a clean new plastic bag (food-grade World Star 1 mil LD bags, or the equivalent, ...), cut slightly larger than the ulcer will be gently conformed to the moist wound contours and sealed onto the zinc oxide paste. The bag will be fenestrated with a small slit using a number 11 scalpel or clean scissors prior to placing it on the ulcer in order to allow excess fluid to escape. The edges of the slit will be approximated. Clean gauze will be placed lightly over the slit to capture escaping fluid. One wrap of stretch gauze will hold the dressing in place. Patients will be instructed to change the dressings daily, irrigating with normal saline at each dressing change.
  Improvised dressing: A piece of a new food-grade plastic bag, cut slightly larger than the ulcer, will be placed over the ulcer, sealed at the edges with an emollient to create an occlusive dressing. The dressing will be gently conformed to the ulcer contours to eliminate dead space, and a slit will be cut in the center to allow excess fluid to escape into a clean absorbent material placed over the slit. The device will be held in place with a wrap of stretch gauze. Ulcers will be rinsed with saline at daily dressing changes, which will be conducted by the patient after they master the procedure.
- Total: Total of all reporting groups
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control) | Total
Number analyzed (Participants) | 16 | 13 | 11 | 40
Age, Continuous [Mean (Full Range); unit: years] | 37.4 [23 to 49] | 44.2 [25 to 61] | 47.9 [29 to 64] | 42.15 [23 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 6 | 16
  Male | 9 | 10 | 5 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Jamaicans of West African descent | 16 | 13 | 11 | 40
Region of Enrollment [Number; unit: participants]
  Jamaica | 16 | 13 | 11 | 40
Initial age of open Sickle Cell Leg Ulcer (SCLU), in weeks [Mean (Full Range); unit: weeks] | 402 [5 to 1560] | 438 [17 to 2040] | 363 [6 to 1560] | 403 [5 to 2040]
Initial depth of study SCLU [Mean (Full Range); unit: millimeters] | 3.94 [1 to 9] | 5.54 [2 to 10] | 4.09 [1 to 8] | 4.50 [1 to 10]
Initial area of study SCLU [Mean (Full Range); unit: centimeters squared] | 43 [0.9 to 198] | 50.7 [1.7 to 304] | 42 [1.2 to 158] | 45.2 [0.9 to 304]
Mid-arm circumference indicates moderate malnutrition [Count of Participants; unit: Participants] — Mid-Upper Arm Circumference is a widely used screening tool for malnutrition. Studies of a black sub-population in South Africa came to the same conclusion as a worldwide USAID study, which found that "MUAC is "highly discriminatory in its ability to distinguish" between individuals with a BMI above or below 18.5kg/m2." Both sets of researchers recommended a MUAC cutoff of ≤ 24.0cm for screening for malnutrition. Counts are given for the number of participants in each group whose MUAC was ≤ 24.0cm.
  Participants | 7 | 2 | 6 | 15
Initial Wound Quality of Life Scores [Mean (Full Range); unit: units on a scale] — The 17 question "Wound-QoL" tool is a questionnaire on Health-related Quality of Life in Chronic Wounds | Version English (US) | Augustin et al. 2014; Blome et al. 2014. Cronbach's alpha between 0.71 and 0.91 and significant convergent validity (r = 0.48 to 0.69). Most participants completed the simple forms on their own each week. Nurses asked participants who did not read well the WQoL questions over the phone. Scores range from 0 to 68. Lower scores indicate better quality of life with respect to the participant's wound.
  units on a scale | 29.875 [5 to 61] | 41.385 [22 to 63] | 42.45 [6 to 63] | 40.825 [5 to 63]
ASCQ-Me baseline scores [Mean (Full Range); unit: units on a scale] — The Adult Sickle Cell Quality of Life Measurement Information System (ASCQ-Me; www.HealthMeasures.net/ASCQ-Me) paper & pencil questionnaire has 5 questions in each of 5 domains answered weekly, plus 14 initial health history questions. Health history raw scores range from 0 - 42, with lower scores indicating a less severe condition. Each weekly domain score is 5 to 25, for a range of 25 - 125; higher scores indicate better sickle-cell related quality of life. Weekly raw scores (not t-scores) are reported here. Nurses asked participants who did not read well the ASCQ-Me questions verbally.
  units on a scale
    Baseline ASCQ-Me Sickle-Cell Related Health History Scores (higher is worse) | 19.9 [1 to 30] | 23.8 [1 to 30] | 19.3 [8 to 30] | 21.0 [1 to 30]
    Baseline ASCQ-Me weekly domain score totals (raw scores, not converted to t-scores) (Lower is Worse) | 85.2 [56 to 119] | 82.4 [38 to 110] | 78.0 [45 to 121] | 82.3 [38 to 121]
Social isolation (lives alone without nearby support) [Count of Participants; unit: Participants] | 1 | 1 | 1 | 3
Use of nicotine (e.g., smoking) in past week (yes/no) [Count of Participants; unit: Participants] — Number of participants who used nicotine (e.g., smoked) in past week.
  Participants | 3 | 2 | 2 | 7
Education level, in years [Mean (Full Range); unit: years] | 11 [6 to 13] | 11 [9 to 16] | 9 [2 to 12] | 10.3 [2 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Wound Complication (A Measure of Dressing Safety)
Description: If wound infection, healing impairing maceration, wound deterioration, etc. are suspected by the patient, the two blinded off-site observers viewing wound photos, or a member of the research study team, all dressings will be removed and the ulcer will be evaluated by a blinded to treatment group member of the medical staff at UHWI who is not involved in the study. Patients and families will be instructed to report any delayed complications, such as wound recurrence, noted within 3 months of study completion. All observed complications were mild pseudomonas infections, and all resolved with the application of dilute vinegar for fewer than two weeks.
Time Frame: During the intervention, potential complications were assessed for presence at least weekly for 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
Participants | 4 | 0 | 0

2. Primary Outcome: Number of Participants Whose Wound Surface Area Decreased (A Measure of Effectiveness)
Description: Subtract the initial wound surface area from the final wound surface area. If the result is a positive number, the wound size remained the same or increased. If the number is negative, the wound size decreased. This is a dichotomous outcome.
Time Frame: Measured at baseline and at 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
Participants | 7 | 10 | 9

3. Primary Outcome: Reported Cultural Acceptability of Available Technology (Improvised) Dressings
Description: Acceptable was defined in the study proposal as an average score of > 4.0
  Question: Does the study dressing's unconventional nature make it unacceptable to you? 5 point Likert scale (higher scores indicate increased acceptability):
  5 - it is not a problem at all 4 - it is an unimportant problem 3 - it is a concern 2 - it is a serious problem
  1 - it is so much of a problem that I would not use it
Time Frame: At final study visit, which took place after approximately 12 weeks of study participation.
Population: In addition to the study participants, the protocol required every family member and study team member who was involved in a participant's wound care to be asked the cultural acceptability question. Only 6 study participants had an involved family member, of whom 5 answered the acceptability question (one declined). In addition, 4 study team members participated in wound care and answered. The PI did not answer because as the developer of the improvised dressing, she has a conflict of interest.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Involved Family Members: Family member who has had some involvement with caring for the participant's wound.
  Maximum of one family member per participant. Surprisingly few family members were willing to have anything at all to do with the participants' wounds. Most either refused to even look at the wounds, or participants hid their wounds from them.
- Involved Health Care Professional (Study Team Member): Due to the COVID-19 pandemic restrictions, many of the health care providers who expected to assist with the study were unable to do so.
  All of the team members who were actively involved in the wound dressing change process participated in the Acceptability question except for the PI, who abstained due to bias in favor of the dressing technique she developed.
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control) | Involved Family Members | Involved Health Care Professional (Study Team Member)
Number analyzed (Participants) | 16 | 13 | 11 | 5 | 4
score on a scale | 4.75 [3 to 5] | 5.0 [5 to 5] | 4.27 [3 to 5] | 4.6 [3 to 5] | 4.25 [3 to 5]

4. Primary Outcome: Change in Patient Overall Quality of Life: ASCQ-Me Questionnaire
Description: The Adult Sickle Cell Quality of Life Measurement Information System tool (ASCQ-Me) Emotional, Pain, Social Functioning, Stiffness, and Sleep Impact Short Forms were administered by interview or self-administered (pencil & paper). Each of these 5 forms is scored from 5 to 25, for a minimum of 25 and maximum of 125 total score. Higher scores indicate better self-reported overall sickle-cell disease-related health. (see Limitations)
  The tool developers expect results to be compared with a reference population whose T scores are provided in their guidance, but only the raw scores are reported here. Also, only the change in the means, from baseline to week 12 (the final scores), for the sum of the five parameters is reported here. This simple calculation does not account for outliers. A more detailed analysis can be requested from the researchers.
Time Frame: Measured at baseline and weekly during the intervention, for 12 weeks. However, the change calculated here is only the difference between baseline and final (week 12) scores for the 5 parameters. Positive differences indicate improved scores.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
score on a scale | 7.516 [-6 to 33] | 4.442 [-19 to 39] | 15.045 [-10 to 42]

5. Secondary Outcome: Percent Change in Wound Surface Area From Baseline (A Measure of Effectiveness)
Description: Measured in cm2 electronically using software that automatically corrects for skew (HealthEPix). Due to the large number of study Sickle Cell Leg Ulcers that were at least partially circumferential, it was not possible to measure the wounds directly from photographs. The wound outlines were traced onto transparent plastic initially and at week 12. These tracings were measured using HealthEPix software, which also computed the wound surface area. The percent change in area was then calculated for each participant using Microsoft Excel (negative = improved). Because tracings were only collected initially and at week 12, it was not possible to obtain weekly ulcer size data. However, HealthEPix did provide accurate wound measurements (including area) from the tracings to allow an accurate calculation of the net change in wound surface area, from which percentage change was calculated. A negative number indicates the ulcer decreased in size.
Time Frame: Measured at baseline and at the conclusion of the study, which is week 12.
Measure: Mean (Standard Deviation); unit: % change in area
Groups:
- Improvised Dressings (Experimental): After initial cleansing/debriding, patients in the improvised dressing group (2) will then have a thin layer zinc oxide paste applied to the dried periwound, carefully avoiding the open wound. A piece of a clean new plastic bag (food-grade World Star 1 mil LD bags, or the equivalent...), cut slightly larger than the ulcer will be gently conformed to the moist wound contours and sealed onto the zinc oxide paste. The bag will be fenestrated with a small slit using a number 11 scalpel or clean scissors prior to placing it on the ulcer in order to allow excess fluid to escape. The edges of the slit will be approximated. Clean gauze will be placed lightly over the slit to capture escaping fluid. One wrap of stretch gauze will hold the dressing in place. Patients will be instructed to change the dressings daily, irrigating with normal saline at each dressing change.
  Improvised dressing: A piece of a new food-grade plastic bag, cut slightly larger than the ulcer, will be placed over the ulcer, sealed at the edges with an emollient to create an occlusive dressing. The dressing will be gently conformed to the ulcer contours to eliminate dead space, and a slit will be cut in the center to allow excess fluid to escape into a clean absorbent material placed over the slit. The device will be held in place with a wrap of stretch gauze. Ulcers will be rinsed with saline at daily dressing changes, which will be conducted by the patient after they master the procedure.
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
% change in area | -1.647 (59.184) | -25.808 (23.628) | -36.071 (44.465)

6. Secondary Outcome: Number of Participants Whose Wound Closed in 12 Weeks
Description: Closed wound - 100% epithelialized with no discernible scab or exudate production (paper napkin remains dry when lightly pressed against area, and no recurrence in the subsequent two weeks), tested by a blinded UHWI physician (not a member of the study team). This outcome measure was modified from "wound closure time from initial assessment " because, due to the pandemic restrictions, participants were rarely able to come for closure verification on the exact week they appeared closed. No ulcers appeared closed before the final three weeks of the study. Two closures were verified on week 11 (group 1 and group 3) and one on week 12 (group 3). All were verified closed at 2 weeks - there were no instances of immediate recurrence.
Time Frame: Assessed Weekly. Closed by the end of the 12 week study period, or not closed by the end of the 12 week period. Verified 2 weeks later. This is a dichotomous variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
Participants | 1 | 0 | 2

7. Secondary Outcome: Choice of Dressings After Study Completion (Which is a Proxy Measure for Dressing Acceptability)
Description: At the conclusion of the study, each participant was given a large quantity of dressing supplies from their choice of the three study protocols as a parting gift. The advanced dressings were unavailable in Jamaica outside of the study, and were the most expensive. The least expensive option was the study dressing (improvised) technique. The usual practice dressings were mid-range in cost and were the most familiar. Most of the participants had a long history of SCLUs (mean age of study ulcer was >7 years), and these ulcers tend to recur, so they expected to require dressings for years to come.
Time Frame: At final study visit, which took place after approximately 12 weeks of study participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
Participants
  Chose usual practice supplies | 2 | 1 | 2
  Chose improvised dressing supplies | 5 | 8 | 3
  Chose advanced dressing supplies | 9 | 4 | 6
  Number who kept same dressings | 2 | 8 | 6

8. Secondary Outcome: Total Materials Costs in US Dollars
Description: Lowest retail costs on Amazon.com were used for donated items, with actual costs for all other dressing materials. Often, participants did not limit the supply counts to those used on their study ulcer, providing instead a weekly total of all supplies used for all of their SCLUs (participants had 1 - 4 SCLUs). When weekly data was missing, it was extrapolated from data in adjacent weeks in which data was provided. Two participants (both in the usual practice group) did not provide any cost data.
Time Frame: During the intervention, measured weekly for 12 weeks. Results were totaled for the entire study duration (12 weeks).
Measure: Mean (Full Range); unit: US Dollars
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 14 | 13 | 11
US Dollars | 108.354 [7.28 to 556.56] | 55.76 [12.12 to 149.69] | 574.15 [81.81 to 2277.72]

9. Secondary Outcome: Average Number of Minutes/Week Spent Performing All Dressing Changes
Description: Estimated by each participant, in minutes, and recorded daily on a data sheet which they submitted weekly. Many participants included the time spent dressing all of their SCLUs, rather than only the study ulcer. The total number of minutes was tallied for each participant for each week. Weekly means were calculated for each participant and then for each group. The range is the range of the participant weekly means.
Time Frame: During the intervention, measured daily for all 12 weeks.
Measure: Mean (Full Range); unit: minutes/week
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 15 | 13 | 11
minutes/week | 153.356 [21.583 to 415] | 144.177 [21 to 266.5] | 86.497 [17.5 to 219]

10. Secondary Outcome: Change in Persistent Wound Pain: Faces Pain Scale - Revised (FPS-R)
Description: Persistent wound pain is wound pain that is present throughout the day, measured using the Faces Pain Scale - Revised (FPS-R), a 0 - 10 scale with 0 being the most desirable outcome. When daily data was missing, blanks were replaced with the average from the other days in the week. The means of scores from the final study week were subtracted from the means of scores from the initial study week, so if the change was an improvement, the value will be a positive number.
Time Frame: Scores were recorded by the participants daily throughout the study. Week 1 means were compared with week 12 means.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
score on a scale | 4.314 [0.11 to 8.26] | 2.469 [.02 to 7.23] | 3.36 [0 to 6.54]

11. Secondary Outcome: Procedural (Dressing Change) Wound Pain: Faces Pain Scale - Revised (FPS-R)
Description: Pain that is the direct result of dressing changes, measured using the Faces Pain Scale - Revised (FPS-R), a 0 - 10 scale with 0 being the most desirable outcome. When daily data was missing, blanks were replaced with the average from the other days in the week. The means of scores from the final study week were subtracted from the means of scores from the initial study week, so if the change was an improvement, the value will be a positive number.
Time Frame: Scores were recorded by the participants daily throughout the study. Week 1 means were compared with week 12 means.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 15 | 13 | 11
score on a scale | 4.23 [0 to 8.4] | 2.61 [0 to 7.21] | 3.00 [0 to 6.32]

12. Secondary Outcome: Change in Patient Wound-specific Quality of Life: Wound-QoL Questionnaire
Description: Assessed with the Wound-QoL tool, a self-assessment tool with 17 questions graded from 0 - 4, with 0 being the most desirable average outcome and 4 being the worst possible average outcome. Possible total scores range from 0 to 68. Sub-scales (body, psyche, and everyday life) can be evaluated independently (contact the researchers about obtaining that data, or for obtaining the weekly raw scores). Higher scores indicate worse SCLU-related quality of life. Final (week 12) total scores were subtracted from baseline total scores to calculate change in scores. If the change was an improvement, the number will be positive. Means for each group are given here.
Time Frame: Measured at baseline and weekly during the intervention, for 12 weeks. Only the change between the baseline score and the week 12 score is reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 16 | 13 | 11
score on a scale | 13.625 [-19 to 38] | 7.692 [-23 to 36] | 15.364 [-20 to 53]

13. Secondary Outcome: Mean Number of Hours/Day the Wound Was Dependent
Description: Approximate amount of time spent standing, or sitting with leg dependent without compression (mean of total hours per day). When daily data was missing, blanks were replaced with the average from the other days in the week. When an entire week was skipped, that participant's week was omitted from the calculations. The means of the daily means for each week for each participant for each group are reported here. Keeping the affected leg elevated when not using compression has been shown to dramatically improve SCLU healing. Therefore, a higher score on this outcome measure could be expected to lead to worse SCLU outcomes.
Time Frame: During the intervention, recorded daily on the participants' weekly data sheet for the entire 12 week study period.
Measure: Mean (Full Range); unit: hours/day
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
Number analyzed (Participants) | 15 | 13 | 11
hours/day | 6.808 [0 to 14.22] | 5.41 [0 to 14.00] | 7.036 [0 to 12.96]

ADVERSE EVENTS:
Time Frame: During the 12 week study period for each participant.
Description: Blinded off site observers and the research team observed photos of wounds weekly and participants were advised to come in for an evaluation if there was any evidence of infection or healing-delaying maceration. Wounds were also assessed in person every 4 weeks.
Arm/Group | Usual Practice (Negative Control) | Improvised Dressings (Experimental) | Advanced Dressings (Positive Control)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 4/16 | 0/13 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Practice (Negative Control) (N=16) | Improvised Dressings (Experimental) (N=13) | Advanced Dressings (Positive Control) (N=11)
Minor Pseudomonas infection (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) — Minor pseudomonas infection in chronic sickle cell leg ulcer. Potential for this adverse event was anticipated in the study protocol and it was quickly managed using the preplanned intervention (dilute vinegar) in all 4 instances.

LIMITATIONS AND CAVEATS:
Due to the pandemic, clinicians hesitated to ask high-risk individuals (sickle cell) to leave home, skewing the sample towards larger, more chronic ulcers in people with poor health overall. A sudden institution of strict movement restrictions led to an abrupt halt to recruitment, transportation shortages, negative interactions with police, and even hunger. Background quality of life deteriorated. Participants had difficulty obtaining pain medications; medication reports were often unreliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04479618/Prot_SAP_ICF_001.pdf